CLINICAL TRIAL: NCT00672789
Title: Adherence to Hydroxyurea in Children With Sickle Cell Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00000118
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2012-11

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle cell anemia; Children; Hydroxyurea; Treatment Adherence
MeSH Terms: conditions — Anemia, Sickle Cell; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Blood Smear Education
  Interventions: Behavioral: Blood smear education
- 2 (Active Comparator): Standard education
  Interventions: Other: standard education

INTERVENTIONS:
Behavioral: Blood smear education — education at baseline and three month follow-up
  Arms: 1
Other: standard education — standard education
  Arms: 2

SUMMARY:
Medication non-adherence is a true public health problem. Despite advancements in the molecular understanding of disease and improvements in therapy, patient health outcomes will not improve unless patients take prescribed medications regularly. Decreasing the gap between efficacious and effective therapy for patients with SCD is an essential research agenda. Hydroxyurea has been shown to be safe and efficacious in children and infants. However, the effectiveness of the prophylaxis depends on adherence to the recommended regimen. Medication adherence in SCD has previously been found to be sub-optimal in patients taking penicillin, desferoxamine, and pain medication. Adherence to HU has been studied to some extent in children with SCD. Based on estimates of adherence in other chronic illness we expect approximately 50% of patients to be >80% adherent with their HU administration. There is no gold standard for improving adherence to treatment. There have been a few attempts in the SCD population to improve adherence. These include a day camp to promote education about desferoxamine and peer support, a combination of a slide-show about SCD and it complications, weekly phone calls by the clinic social worker and a calendar, and a seven-phase educational program. Given the striking improvements in the peripheral blood smear findings of patients with SCD on HU therapy, with reduction in the numbers of sickled cells, we hypothesize that viewing the peripheral blood smear of patients with poor adherence to HU compared to a blood smear of someone on HU can be used to improve adherence in non-adherent patients.

We will conduct a randomized trial between the intervention of regularly showing children and their parents the peripheral blood smear and standard care, including reminders of the importance of compliance and review of complete blood count parameters, including WBC, MCV, and Hgb concentration. The outcome measures will be increase in hemoglobin concentration and %HbF and increase in perceived QOL. QOL will be measured with age-appropriate and parent/proxy PedsQL™. Medication adherence will also be monitored throughout the study with pharmacy prescription refills, physician assessment, and self-report via a visual analogue scale. Adherence estimates, hemoglobin concentration, %HbF and QOL will be measured at baseline, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell anemia
* on Hydroxyurea for at least six months
* age 2-17.9 years

Exclusion Criteria:

* none

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
treatment adherence | six months

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Thornburg, MD, MS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States